CLINICAL TRIAL: NCT00989651
Title: A Phase I Study of Intravenous Carboplatin/Paclitaxel or Intravenous and Intraperitoneal Paclitaxel/Cisplatin in Combination With Continuous or Intermittent /CTEP-Supplied Agent ABT-888 (NSC #737664) and CTEP-Supplied Agent Bevacizumab (NSC #704865) in Newly Diagnosed Patients With Previously Untreated Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Carboplatin, Paclitaxel, Bevacizumab, and Veliparib in Treating Patients With Newly Diagnosed Stage II-IV Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03730; NCI-2011-03730 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-9923; CDR0000656038; GOG-9923 (Other: NRG Oncology); GOG-9923 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Fallopian Tube Carcinoma; Fallopian Tube Carcinosarcoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Neoplasm; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Ovarian Brenner Tumor; Ovarian Carcinoma; Ovarian Carcinosarcoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Tumor; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIA Ovarian Cancer AJCC V6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Ovarian Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Ovarian Cancer AJCC v6 and v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms; Brenner Tumor; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen I (paclitaxel, carboplatin, bevacizumab, veliparib) (Experimental): Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes (beginning in course 2) on day 1. Patients also receive veliparib PO BID on days 1-21. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment with bevacizumab repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Veliparib
- Regimen II (paclitaxel, carboplatin, bevacizumab, veliparib) (Experimental): Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Patients also receive carboplatin, bevacizumab, and veliparib as in Regimen I. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment with bevacizumab repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Veliparib
- Regimen III (paclitaxel, cisplatin, bevacizumab, veliparib) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1 and IP on day 8, and cisplatin IP on day 1 or 2. Patients also receive bevacizumab and veliparib as in Regimen I. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Veliparib

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Regimen I (paclitaxel, carboplatin, bevacizumab, veliparib); Regimen II (paclitaxel, carboplatin, bevacizumab, veliparib)
Drug: Cisplatin — Given IP
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Regimen III (paclitaxel, cisplatin, bevacizumab, veliparib)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV or IP
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with carboplatin, paclitaxel, and bevacizumab in treating patients with newly diagnosed stage II-IV ovarian epithelial, fallopian tube, or primary peritoneal cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cells to repair themselves from damage and survive. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab, a type of drug called a monoclonal antibody, blocks tumor growth by targeting certain cells and preventing the growth of new blood vessels that tumors need to grow. Giving veliparib together with carboplatin, paclitaxel, and bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose-limiting toxicities of ABT-888 (veliparib) when administered using continuous versus intermittent dosing schedules with intravenous carboplatin, paclitaxel and bevacizumab using two different treatment regimens; or with intraperitoneal cisplatin and intravenous and intraperitoneal paclitaxel and bevacizumab in women with newly diagnosed, previously untreated, epithelial ovarian, fallopian tube, or primary peritoneal cancer.

II. To determine the feasibility of these treatment regimens over four cycles in a 2-stage group sequential design once the MTD is established.

III. To assess the toxicity of these regimens using Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. To estimate the response rate (in measurable disease patients) and progression-free survival in patients treated with these treatment regimens.

TERTIARY OBJECTIVES:

I. To assess the extent of poly-ADP-ribose polymerase (PARP) inhibition in peripheral blood mononuclear cells (PBMCs) on day 1 of cycles 1 and 2.

II. To assess genomic breast cancer, early onset (BRCA) mutation status in all patients in regimens I and II with continuous ABT-888 dosing and descriptively correlate with toxicity and efficacy.

OUTLINE: This is a dose-escalation study of veliparib followed by a feasibility study. Patients are sequentially assigned to 1 of 3 treatment regimens.

REGIMEN I: Patients receive paclitaxel intravenously (IV) over 3 hours, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes (beginning in course 2) on day 1. Patients also receive veliparib orally (PO) twice daily (BID) on days 1-21. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment with bevacizumab repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.

REGIMEN II: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15. Patients also receive carboplatin, bevacizumab, and veliparib as in Regimen I. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment with bevacizumab repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.

REGIMEN III: Patients receive paclitaxel IV over 3 hours on day 1 and intraperitoneally (IP) on day 8, and cisplatin IP on day 1 or 2. Patients also receive bevacizumab and veliparib as in Regimen I. Treatment repeats every 21 days for 6 courses. Patients then receive bevacizumab alone on day 1. Treatment repeats every 21 days for 16 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, or carcinosarcoma stage II, III, or IV with either optimal (=< 1 cm residual disease) or suboptimal residual disease
* All patients must have a procedure for determining diagnosis of epithelial ovarian, fallopian tube, primary peritoneal, or carcinosarcoma with appropriate tissue for histologic evaluation
* Patients with the following histologic cell types are eligible:

  * Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial adenocarcinoma, transitional cell carcinoma, malignant Brenner's tumor, adenocarcinoma not otherwise specified (N.O.S.) or carcinosarcoma
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, equivalent to CTEP Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, grade 1; this ANC cannot have been induced or supported by granulocyte colony stimulating factors
* Platelets greater than or equal to 100,000/mm^3
* Regimens I and II: Creatinine =< 1.5 x institutional upper limit normal (ULN), CTCAE grade 1

  * Regimen III: Creatinine no greater than the institutional upper limits of normal
* Bilirubin less than or equal to 1.5 x ULN (CTEP CTCAE version 4.0, grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3 x ULN (CTEP CTCAE version 4.0, grade 1)
* Alkaline phosphatase less than or equal to 2.5 x ULN (CTEP CTCAE version 4.0, grade 1)
* Albumin greater than or equal to 3.0 g/dL
* Neuropathy (sensory and motor) less than or equal to CTEP CTCAE version 4.0, grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) < 1.5 x ULN
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Patients must be entered between 1 and 12 weeks after initial surgery performed for the combined purpose of diagnosis, staging and cytoreduction
* Patients who have met the pre-entry requirements specified
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with a current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent invasive epithelial ovarian, primary peritoneal or fallopian tube cancer treated with surgery only (such as patients with stage IA or IB low-grade epithelial ovarian or fallopian tube cancers) are not eligible

  * NOTE: Patients with a prior diagnosis of a borderline tumor that was surgically resected and who subsequently develop an unrelated, new invasive epithelial ovarian, peritoneal primary or fallopian tube cancer are eligible, provided that they have not received prior chemotherapy for any ovarian tumor
* Patients with synchronous primary endometrial cancer or a past history of endometrial cancer, unless all of the following conditions are met:

  * Stage not greater than IB
  * No more than superficial myometrial invasion
  * No vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor within the last five years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with acute hepatitis or active infection that requires parenteral antibiotics
* Patients with serious non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days; patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures or history of seizures, and/or any CNS metastases are ineligible
* Patients with history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study are ineligible
* Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg
* Myocardial infarction or unstable angina < 6 months prior to registration
* New York Heart Association (NYHA) class II or higher congestive heart failure
* Serious cardiac arrhythmia requiring medication
* CTEP CTCAE version 4.0, grade 2 or higher peripheral ischemia (brief [< 24 hours (hrs)] episode of ischemia managed non-surgically and without permanent deficit)
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Patients with clinically significant proteinuria (urine protein creatinine ratio greater or equal to 1.0)
* Patients with invasive procedures or anticipation of invasive procedures within the following timeframes as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab therapy (cycle 2)
  * Major surgical procedure anticipated during the course of the study
  * Core biopsy within 7 days prior to the first date of bevacizumab therapy (cycle 2)
* Patients who are pregnant or nursing
* Patients with clinical symptoms or signs of gastrointestinal obstruction and who require parenteral hydration or nutrition
* Patients with GOG performance status of 3 or 4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2009-10-28 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) occurring in the first or second course of treatment (dose-escalation phase) | Up to day 42
Incidence of DLTs occurring in the first 4 courses of treatment (feasibility phase) | Up to day 84

SECONDARY OUTCOMES:
Objective tumor response (complete and partial response) as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 11 years
  Tabulated by regimen and BRCA mutation status.
Progression-free survival | Time from start of treatment to time of progression or death, assessed up to 11 years
  Summarized using Kaplan-Meier plots by BRCA mutation status.
Incidence of toxicity, graded according to National Cancer Institute CTCAE version 4.0 | Up to 30 days after last dose of treatment
  Tabulated by regimen and by BRCA mutation status.

OTHER OUTCOMES:
Change in PARP inhibition in PBMCs | Day 1 to day 22 (day 1 of course 1 to day 1 of course 2)
  PARP inhibition in PBMCs in each course (courses 1 and 2) and the change from course1 to course 2 will be summarized by dose level and regimen using descriptive statistics (e.g., mean, standard deviation, median, quartiles) and using graphs. In addition, linear models may be used to assess the association between PARP inhibition and dose level with transformations of the PARP inhibition as appropriate.
Genomic BRCA mutation status | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Bell-McGuinn, Principal Investigator — NRG Oncology
Locations (23):
- United States (23):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Colorado Hospital, Aurora, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Gillen J, Miller A, Bell-McGuinn KM, Schilder RJ, Walker JL, Mathews CA, Duska LR, Guntupalli SR, O'Cearbhaill R, Hays J, Hagemann AR, Gray HJ, Gordon SW, Armstrong DK, Chen A, Fracasso PM, Aghajanian C, Moore KN. Post hoc analyses of GOG 9923: Does BRCA status affect toxicities?: An NRG oncology study. Gynecol Oncol. 2021 May;161(2):512-515. doi: 10.1016/j.ygyno.2021.01.037. Epub 2021 Feb 17. PMID 33610319
- [Derived] Moore KN, Miller A, Bell-McGuinn KM, Schilder RJ, Walker JL, O'Cearbhaill RE, Guntupalli SR, Armstrong DK, Hagemann AR, Gray HJ, Duska LR, Mathews CA, Chen A, O'Malley D, Gordon S, Fracasso PM, Aghajanian C. A phase I study of intravenous or intraperitoneal platinum based chemotherapy in combination with veliparib and bevacizumab in newly diagnosed ovarian, primary peritoneal and fallopian tube cancer. Gynecol Oncol. 2020 Jan;156(1):13-22. doi: 10.1016/j.ygyno.2019.10.012. Epub 2019 Nov 7. PMID 31708167